CLINICAL TRIAL: NCT05351086
Title: A Double Dummy, Double-blind Study to Assess the Safety, Tolerability, and Pharmacokinetics of PUR3100 in Health Adults
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of PUR3100 in Health Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmatrix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 601-0022
Record Dates: First submitted 2022-04-19; First posted 2022-04-28 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Healthy
MeSH Terms: interventions — Dihydroergotamine

STUDY DESIGN:
Intervention Model Description: Double Dummy, Double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A computerized randomization scheme will be created and shall be considered blinded (as per the following). The randomization is available only to the clinical research unit pharmacy staff that are preparing the drug who will not be involved in any other aspect of the study including administration of the drug. It will not be made available to the subjects, site PI, or members of the staff responsible for the monitoring and evaluation of study assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Inhaled placebo and IV D.H.E. 45 1 mg (Experimental)
  Interventions: Drug: Dihydroergotamine (D.H.E 45); Other: Matching Placebo for PUR3100
- Inhaled PUR3100 0.5 mg and IV placebo (Experimental)
  Interventions: Drug: PUR3100; Other: Matching Placebo for D.H.E 45
- Inhaled PUR3100 1.0 mg and IV placebo (Experimental)
  Interventions: Drug: PUR3100; Other: Matching Placebo for D.H.E 45
- Inhaled PUR3100 1.5 mg and IV placebo (Experimental)
  Interventions: Drug: PUR3100; Other: Matching Placebo for D.H.E 45

INTERVENTIONS:
Drug: PUR3100 — PUR3100 is an inhalation powder containing DHE, an anti-migraine treatment with broad spectrum agonist activity against 5-hydroxytryptamine (5-HT), dopamine, and adrenergic receptors. PUR3100 is provided as 500 µg dose strength capsules. Each capsule contains the drug substance, DHE mesylate, with mannitol, leucine, and sodium chloride as excipients.
  Arms: Inhaled PUR3100 0.5 mg and IV placebo; Inhaled PUR3100 1.0 mg and IV placebo; Inhaled PUR3100 1.5 mg and IV placebo
Drug: Dihydroergotamine (D.H.E 45) — D.H.E. 45 is ergotamine hydrogenated in the 9, 10 position as the mesylate salt. It is supplied as a clear, colorless solution supplied in sterile ampules for IV, intramuscular, or subcutaneous administration containing (per mL) DHE mesylate, USP 1 mg, ethanol, 94% w/w. 6.2% by volume, glycerin 15% by weight, and water for injection.
  Arms: Inhaled placebo and IV D.H.E. 45 1 mg
Other: Matching Placebo for PUR3100 — Each capsule of matching placebo is filled with iSPERSE powder comprised of mannitol, leucine, and sodium chloride. The PUR3100 inhalation powder is administered using the supplied RS01 inhalation device (RS01 UHR2, Plastiape S.p.A.).
  Arms: Inhaled placebo and IV D.H.E. 45 1 mg
Other: Matching Placebo for D.H.E 45 — The matching placebo for D.H.E. 45 is 0.9% sterile saline for injection.
  Arms: Inhaled PUR3100 0.5 mg and IV placebo; Inhaled PUR3100 1.0 mg and IV placebo; Inhaled PUR3100 1.5 mg and IV placebo

SUMMARY:
A Double Dummy, Double-blind Study to Assess the Safety, Tolerability, and Pharmacokinetics of PUR3100 in Healthy Adults

DETAILED DESCRIPTION:
This is a randomized, parallel group, double-blind, double dummy study.

Following screening and confirmation of eligibility, twenty-four healthy subjects will be evenly randomized to 1 of the 4 dose groups of 6 subjects each. Subjects will receive intravenous (IV) dihydroergotamine (D.H.E) or IV placebo and dry powder inhalation of 0.5mg of PUR3100, 1.0 mg of PUR 3100, 1.5 mg of PUR 3100, or placebo.

All potential subjects will complete screening between 28 days and 2 days prior to study unit check-in on Day -1. Subjects will remain in the study unit for 3 days post check-in and will be dosed each day at the study site.

A follow up visit will occur 4 days after the last dose of study drug, on Day 7 of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 to 55 years of age with a body mass index ≥17 and ≤35 kg/m2.
2. Subject has normal screening and baseline blood pressure, defined as a systolic value ≥90 mmHg and ≤140 mmHg and a diastolic value >60 mmHg and <90 mmHg.
3. Female subjects who are of childbearing potential and male subjects with female partner(s) of childbearing potential must agree to use an effective contraceptive throughout the study (e.g., oral contraceptives or Norplant®; a reliable double barrier method of birth control [diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam]; intrauterine devices; partner with vasectomy; or abstinence) and for at least 90 days after study drug administration. In addition, female subjects must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to dosing. Note: Women of non-childbearing potential may be enrolled if they are:

   1. Surgically sterile (e.g., hysterectomy with or without oophorectomy; fallopian tube ligation; endometrial ablation), for at least 30 days prior to signing the ICF
   2. Post-menopausal (≥ 12 consecutive months of spontaneous amenorrhea and > 50 years of age)
4. Female subjects must agree not to donate ova/oocytes during the study and for 90 days after the last dose of IMP.
5. Male subject must agree not to donate semen during the study and for 90 days after the last dose of IMP.
6. Subject is able and willing to abstain from alcohol for 48 hours prior to admission to the study unit and throughout the entire study until completion of the Day 7 follow up visit.
7. Subject is willing to participate in the study, comply with the study requirements, and voluntarily provide written informed consent.
8. Subject can read, write, and speak English.
9. Subject is mentally competent to provide informed consent.
10. Subject can perform technically acceptable spirometry at screening.
11. Subject can demonstrate the correct inhalation technique for use of the delivery device and to generate sufficient peak inspiratory flow (PIF) of at least 40 L/min using the In-Check DIAL device at screening.

Exclusion Criteria:

1. Subject has a history of proven or suspected coronary artery disease (CAD), coronary vasospasm (including Prinzmetal's angina), peripheral vascular disease, or other ischemic diseases (e.g., ischemic bowel syndrome or Raynaud's syndrome) or cardiac disorder (e.g., any clinically significant dysrhythmia), any history of heart attack or stroke, hypertension, diabetes mellitus, liver or kidney disease, aortic aneurysm, chronic pulmonary disease, or recent (within 3 months) sepsis or vascular surgery.
2. Subject has a current diagnosis of asthma, chronic obstructive pulmonary disease, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, interstitial lung disease, known alpha-1 antitrypsin deficiency, or other active pulmonary disease.
3. Subject has clinically significant abnormal laboratory values at screening that, in the opinion of the investigator would make the subject inappropriate for the study or put the subject at undue risk, specifically liver function tests (LFTs) >1.5 times the upper limit of normal (ULN); hemoglobin <10 gm/dL; absolute neutrophil count (ANC) <2.0 x 109/L; white blood cells (WBC) ˃11 x 109/L; platelets <100,000 or >500,000; international normalization ratio (INR) >1.3.
4. Subject has a QTcF of >450 msec in males or >470 msec in females at screening.
5. Subject has forced expiratory volume in 1 second (FEV1) or forced vital capacity (FVC) on screening spirometry that is less than 80% predicted.
6. Subject has a history of illicit drug or alcohol abuse within the past 12 months prior to screening.
7. Subject smokes more than 5 cigarettes per day or vapes more than 5 times per day with devices that deliver nicotine.
8. Subject has a history of nicotine replacement products daily within 6 months prior to screening.
9. Subject has a positive alcohol test result at screening.
10. Subject has a positive urine drug test result at screening, unless the result can be explained by the subject's current medications, in which case the PI should discuss the disposition of the subject with the Sponsor. Cannabidiol (CDB) and tetrahydro cannabinol (THC) use is prohibited.
11. Subject has a known sensitivity to the study drug or any of the excipients of the formulation, or history of clinically significant sensitivity to any agent that, in the opinion of the investigator, would make participation in the study inadvisable.
12. Subject has donated blood or blood products or had substantial loss of blood (more than 500 mL) within 6 weeks prior to screening.
13. Subject has participated in an interventional study involving an experimental therapeutic agent within 3 months of screening.
14. Women who have a positive serum β-human chorionic gonadotropin (hCG) pregnancy test at screening or a positive urinary hCG pregnancy test prior to dosing, is pregnant, lactating, or planning to become pregnant during the study or within 90 days after conclusion of study participation.
15. Subject has a positive hepatitis B surface antigen (HbsAg), hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV) test result. Subjects who are hepatitis B surface (HBs) antibody positive or hepatitis B (HB) core antibody positive are not excluded provided the HBsAg result is negative. Subjects who are HCV antibody positive are not excluded if a subsequent HCV RNA test is negative.
16. Subject has a planned surgery or procedure during participation in the study and for 28 days after the conclusion of study participation.
17. Subject is an employee of the investigator or study site with direct involvement in the proposed study or other studies under the direction of that investigator or study site or is a family member of a study site employee or the investigator.
18. Subject has a current or chronic history of liver disease or known hepatic or biliary abnormalities (except for Gilbert's syndrome or asymptomatic gallstones).
19. The subject is unable or unwilling to comply fully with the study protocol.
20. Subject is mentally or legally incapacitated.
21. Subject is unable or unwilling to undergo multiple venepuncture procedures or the subject has poor access to veins suitable for cannulation.
22. There is a condition or situation that, in the opinion of the investigator, would make participation in the study inadvisable.
23. Subject has a history of chronic uncontrolled disease including, but not limited to, cardiovascular, endocrine, neurological, hepatic, gastrointestinal, renal, hematologic, urologic, immunologic, or ophthalmic diseases that, in the opinion of the investigator, would make participation in the study inadvisable.
24. Subject has had major surgery within 6 weeks prior to screening.
25. Subject has a disclosed history, or one known to the investigator, of significant noncompliance in previous investigational studies or with prescribed medications.
26. Subject requires supplemental oxygen, even on an occasional basis.
27. Subject received a live vaccine within 14 days prior to screening.
28. Caffeine-containing beverage e.g coffee, tea, or caffeine sodas or power drinks (greater than 3 cups per day, 1 cup=250 mL) within 3 months prior to screening. Subject is UN able and unwilling to abstain from tea, coffee, or caffeine-containing beverages for 48 hours prior to admission to the study unit and throughout the entire study until completion of the Day 7 follow up visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Day 1 through Day 3adult subjects
  To determine the safety and tolerability of single doses of inhaled PUR3100 in healthy through the review of AEs
Maximum Plasma Concentration [Cmax] | Day 1 through Day 3
  To characterize the systemic pharmacokinetics (PK) of single doses of inhaled PUR3100 in healthy adult subjects by measuring the maximum drug concentration in blood plasma.
  This will also be compared to Cmax of participants who receive IV D.H.E. 45.
Last Observed Plasma Concentration [Clast] | Day 1 through Day 3
  To characterize the systemic pharmacokinetics (PK) of single doses of inhaled PUR3100 in healthy adult subjects by measuring the last observed quantifiable concentration of PUR 3100 in blood plasma.
  This will also be compared to Clast of participants who receive IV D.H.E. 45.
Time to Peak Drug Concentration [Tmax] | Day 1 through Day 3
  To characterize the systemic pharmacokinetics (PK) of single doses of inhaled PUR3100 in healthy adult subjects by measuring the time time it takes for a drug to reach the maximum concentration (Cmax).
  This will also be compared to Tmax of participants who receive IV D.H.E. 45.
Time of last measurable concentration [Tlast] | Day 1 through Day 3
  To characterize the systemic pharmacokinetics (PK) of single doses of inhaled PUR3100 in healthy adult subjects by measuring the time time it takes for a drug to reach the last measurable concentration of PUR 3100 in blood plasma.
  This will also be compared to Tlast of participants who receive IV D.H.E. 45.
Area under the curve [AUC (0-t), AUC (0-inf), AUC (0-2h)] | Day 1 through Day 3
  To characterize the systemic pharmacokinetics (PK) of single doses of inhaled PUR3100 in healthy adult subjects by measuring the drug concentration in blood plasma over time.
  This will also be compared to the AUC (0-t), AUC (0-inf), and AUC (0-2h) of participants who receive IV D.H.E. 45.
Half Life [ t 1/2 ] | Day 1 through 3
  To characterize the systemic pharmacokinetics (PK) of single doses of inhaled PUR3100 in healthy adult subjects by measuring the time it takes for the amount of drug in the blood to reduce by 50%.
  This will also be compared to the half life of participants who receive IV D.H.E. 45.
Clearance (CL/F) | Day 1 through Day 3
  To characterize the systemic pharmacokinetics (PK) of single doses of inhaled PUR3100 in healthy adult subjects.
  This will also be compared to the CL/F of participants who receive IV D.H.E. 45.
Apparent Volume of Distribution During Terminal Phase (Vz/F) | Day 1 through Day 3
  To characterize the systemic pharmacokinetics (PK) of single doses of inhaled PUR3100 in healthy adult subjects.
  This will also be compared to the Vz/F of participants who receive IV D.H.E. 45.

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Melbourne, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No